CLINICAL TRIAL: NCT03748459
Title: Patient and Observer Graded Rhinoplasty Scar Outcomes: a Randomized-Controlled Trial of Fast Absorbing Versus Permanent Columellar Suture Closure
Brief Title: Rhinoplasty Scar Comparison
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 00066546
Record Dates: First submitted 2018-11-19; First posted 2018-11-20 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Surgical Incision; Nose Deformity
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Permanent suture: Subjects will have skin closure with permanent suture (prolene) (6-0 polypropylene) in open rhinoplasty.
  Interventions: Other: Closure with Permanent Suture
- Resorbable suture: Subjects will have skin closure with Resorbable Suture (5-0 fast absorbing plain gut) in open rhinoplasty
  Interventions: Other: Closure with Resorbable Suture

INTERVENTIONS:
Other: Closure with Permanent Suture — Skin closure with permanent suture (prolene) (6-0 polypropylene) in open rhinoplasty.
  Groups: Permanent suture
Other: Closure with Resorbable Suture — Skin closure with Resorbable Suture (5-0 fast absorbing plain gut) in open rhinoplasty.
  Groups: Resorbable suture

SUMMARY:
Traditional suture closure of the columellar scar in rhinoplasty is achieved with permanent skin sutures. These sutures create less inflammation and are thought to lead to improved final scar outcomes. However, permanent sutures require removal which creates pain and inconvenience for the patient. Some surgeons use fast absorbing sutures that do not require removal. The difference in final scar outcome based on suture material used has not been well studied. This study will examine the final scar outcomes of rhinoplasty incisions sutured with traditional permanent suture compared to fast absorbing suture. If scar outcomes are similar between these groups as judged by the patients and blinded observers, rhinoplasty surgeons may be able to preferentially utilize absorbable sutures for incision closure and avoid the pain and inconvenience for the patient during suture removal

ELIGIBILITY:
Inclusion Criteria

•Adult (age ≥ 18 years) patients undergoing primary open rhinoplasty surgery for any reason with any of the study surgeons.

Exclusion Criteria

* Patients undergoing rhinoplasty for cleft nasal deformity or nasal reconstruction related to cancer resection
* Patients with previous surgery that involved a columellar incision. Patients with history of previous nasal surgery that did not involve an incision on the columella may be included
* Patients with known history of cutaneous disorder that affects scaring such as personal history of keloid formation, collagen vascular disease, or previous radiation to the surgical site
* Inability or unwillingness of subject to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients seeking rhinoplasty surgery with one of the investigators.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Patient Scar Assessment | 12 months after surgery
  Patient scar assessment will be done with a patient completed questionnaire. The questionnaire is a validated scar assessment instrument for self rating of surgical scars by patients for a minimum rating of 28 (best scar) to 112 (worst scar)
Clinician Scar Assessment | 12 months after surgery
  Clinician scar assessment will be done using photographs of the scar 12 months after surgery. Clinicians will use a validated clinician scar grading tool for evaluation of surgical scars with a range of 0 (worst scar) to 5 (best scar)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Ralph Johnson VA Medical Center, Charleston, South Carolina